CLINICAL TRIAL: NCT01913301
Title: A Randomized Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Effects of Alagebrium on Exercise in Subjects With Diastolic Heart Failure
Acronym: BREAK-DHF-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor lost funding
Sponsor: Cardiovascular Clinical Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-711-0530
Record Dates: First submitted 2013-02-15; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-02

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alagebrium (Experimental)
  Interventions: Drug: Alagebrium

INTERVENTIONS:
Drug: Alagebrium

SUMMARY:
The purpose of the study is to gather information regarding the safety and effectiveness of an investigational drug called Alagebrium when used treating Heart Failure in relation to exercise tolerance after 6 months in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 50 years of age or older.
2. Diagnosis of diabetes OR a diagnosis of hypertension requiring therapy.
3. Echocardiographic ejection fraction ≥ 45% verified within 1 year prior to baseline, assuming no intercurrent cardiac event between the echo and screening.
4. Echocardiographic evidence of diastolic dysfunction as defined by an E/E' ≥ 12 determined within 1 year prior to baseline; sinus rhythm required at time of echo.
5. Previous hospitalization due to heart failure OR a current or previous BNP ≥ 100 pg/mL.
6. New York Heart Association (NYHA) functional class II-IV.
7. At least 1 month between hospitalization for heart failure and randomization.
8. Stable doses of heart failure medications (diuretics, ACE inhibitors, ARB's, beta-adrenergic antagonists, aldosterone antagonists) for at least 1 month prior to randomization.
9. Able to understand content of and willing to provide written informed consent.
10. Agree to use adequate contraception during the study if premenopausal. -

Exclusion Criteria:

1. Ejection fraction < 45%.
2. Screening Six-minute walk test > 450 meters or < 100 meters
3. Clinically significant cardiac valvular disease (mitral regurgitation (MR) > grade I, aortic insufficiency (AI) > grade 1, mitral stenosis (MS), aortic stenosis (AS)).
4. History of stroke, any sequelae of a transient ischemic attack (TIA), or reversible ischemic neurological defect (RIND) within 6 months prior to screening.
5. History of acute myocardial infarction within 6 months prior to screening.
6. Severe COPD as defined by O2 or steroid dependence.
7. History of systemic inflammatory or collagen vascular disease.
8. Active and or treated malignancies within 12 months prior to Visit 1 with the exception of basal cell carcinoma.
9. Any significant systemic illness(es) or medical condition(s) that could lead to difficulty complying with the protocol; or any concurrent condition(s) which, in the investigator's opinion, would prohibit the subject from completing the study, or would not be in the best interest of the subject.
10. Estimated glomerular filtration rate (GFR) ≤ 30 mL/min/1.73m² as calculated by Modification of Diet in Renal Disease (MDRD) study equation [MDRD = 186 X serum creatinine (mg/dl) 1.154 X years -0.203 X (0.742 if female) X (1.210 if African American)].
11. Liver function tests (SGOT and/or SGPT) > 2.5 times the upper limit of normal range.
12. Hb < 10 g/dL.
13. Use of any investigational drug(s) within 30 days prior to screening.
14. Previous exposure to alagebrium.
15. Known seropositivity for HIV or hepatitis C, or presence of hepatitis B surface antigen.
16. Pregnancy or active breast-feeding. Urine pregnancy tests will be performed on all women who are not post-menopausal for at least 1 year.

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Exercise Tolerance | Change from baseline at Week 24
  To evaluate the safety and efficacy of alagebrium in subjects diagnosed with diastolic heart failure. The primary variable for assessing efficacy will be assessment of exercise tolerance using the Six-minute walk test.